CLINICAL TRIAL: NCT03827980
Title: LOOP- Long- and Midterm Outcomes of Osteoarticular Infections in Paediatric Patients.
Brief Title: Long- and Midterm Outcomes of Osteoarticular Infections in Paediatric Patients
Acronym: LOOP
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Ulrich Heininger (Other)
Collaborators: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Ulrich Heininger, Chair, Infectious Diseases/Vaccinology, University Children's Hospital Basel
Organization: University Children's Hospital Basel (Other)
Other Study IDs: 2018-02393
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Acute Haematogenous Osteomyelitis; Septic Arthritis
Keywords: Acute Haematogenous Osteomyelitis; Septic Arthritis; Outcome; Osteoarticular Infections; Follow-up
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention, only clinical examination — standardised interview and clinical examination

SUMMARY:
Multi-centre clinical follow-up study on patients with a history of acute haematogenous osteomyelitis and/or septic arthritis. The aim is to describe the frequency of sequelae in these former patients with osteoarticular infections. Patients will be invited to participate in a single follow-up visit including a standardised interview and a clinical examination. The collected data will be analyzed together with data from the patient's hospital stay.

DETAILED DESCRIPTION:
Clinical follow-up study on patients with a history of acute haematogenous osteomyelitis and/or septic arthritis and were admitted to one of the participating centres between 2005 and 2014.

Former patients will be invited to participate in a single-follow-up visit which comprises a standardised interview (pain, disabilities in daily life and regarding sports) and a standardized clinical examination of the previously affected body part. This includes assessment of range of motion in affected and adjacent joints and in case of previously affected lower extremity leg axis, gait and body height (percentile).

The data collected during the follow-up visit will be analyzed in a descriptive manner together with data of the patient's hospital stay including baseline data, laboratory works, microbiological results and both antibiotic and surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were previously admitted to the participating centres between January 2005 and November 2014
* Patients with an International Classification of Disease code (ICD-10) discharge code of acute osteomyelitis (M86.00-M86.99) and/or septic arthritis (M00.00-M00.99)

Exclusion Criteria:

* onset of symptoms > 2 weeks before admission
* history of penetrating wound or Prior surgery at affected limb
* incorrect ICD-10 coding
* chronic or severe underlying disease or Treatment at time of infection that possibly compromises the patient's immunologic Response (e.g. cancer, immunodeficiency, immunosuppressive therapy)
* insufficient command of German language to understand patient Information and informed consent

Ages: 4 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Former patients admitted to one of the participating centres for an acute osteoarticular infection.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
subjective sequelae score of previously affected body region: lower extremity | Day 1 (at single study visit)
  Assessment of current pain and ability to perform physical activities summarized in a Subjective Sequelae Score modified after the PODCI (Pediatric Outcomes Data Collection Instrument) questionnaire and score:
  Lower Extremity: 11 Questions, Points 0-35, 0 = no disabilities, 1-11 = minor disability, 12-23 = moderate disability, 24-35 = severe disability Question 1: Current pain: (0-5 Points: never/less than once a month/once a month/once a week/more than once a week/daily) Questions 2-11 (0-3 Points never/less than once a month/once a month/once a week/more than once a week/daily) 2) Short distance running 3) Long distance running 4) Walking > 100m 5) Walking > 1000m 6) Climbing stairs 7) Walking uphill 8) Walking downhill 9) Participation in ball games/sports 10) Kneeling down 11) Sitting low (e.g. car, couch)
subjective sequelae score of previously affected body region: upper extremity | Day 1 (at single study visit)
  Assessment of current pain and ability to perform physical activities summarized in a Subjective Sequelae Score modified after the PODCI (Pediatric Outcomes Data Collection Instrument) questionnaire and score:
  Upper Extremity: 6 Questions, Points 0-35, 0 = no disabilities, 1-6 = minor disability, 7-13 = moderate disability, 14-20 = severe disability Question 1: Current pain: (0-5 Points: never/less than once a month/once a month/once a week/more than once a week/daily) Questions 2-6 (0-3 Points never/less than once a month/once a month/once a week/more than once a week/daily) 2) Light work with upper body 3) Heavy work (e.g. Lifting heavy things) 4) Using Tools 5) Putting weight on upper body 6) Overhead work
relevant restricted range of motion | Day 1 (at single study visit)
  restricted range of motion of > 20° of previously affected body part / joint compared to the other side

SECONDARY OUTCOMES:
asymmetric axis of leg or arm | Day 1 (at single study visit)
  asymmetric leg or arm axis of previously affected lower or upper limb, respectively.
limb length discrepancy of > 1cm | Day 1 (at single study visit)
  asymmetric length of legs/arms of previously affected lower or upper limb, respectively.
abnormal gait (only in case of previously affected lower limb) | Day 1 (at single study visit)
  abnormal gait (e.g. limping) at examination
z-score decline of body height since hospital discharge (only in case of previously affected lower limb) | variable, between 4 and 14 years, depending on time frame between date of discharge and today's study visit.
  decline in body height between hospital discharge and study visit

CONTACTS AND LOCATIONS:
Overall Officials: Nora Manz, MD, Principal Investigator — University Children's Hospital Basel
Locations (2):
- Switzerland (2):
  - University Children's Hospital Basel, Basel, Canton of Basel-City
  - Children's Hospital Lucerne, Lucerne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manz N, Krieg AH, Heininger U, Ritz N. Evaluation of the current use of imaging modalities and pathogen detection in children with acute osteomyelitis and septic arthritis. Eur J Pediatr. 2018 Jul;177(7):1071-1080. doi: 10.1007/s00431-018-3157-3. Epub 2018 May 4. PMID 29728840
- [Derived] Manz N, Krieg AH, Buettcher M, Ritz N, Heininger U. Long-Term Outcomes of Acute Osteoarticular Infections in Children. Front Pediatr. 2020 Nov 25;8:587740. doi: 10.3389/fped.2020.587740. eCollection 2020. PMID 33335875